CLINICAL TRIAL: NCT00972205
Title: A Pharmacodynamic Study of the P-glycoprotein (Pgp) Antagonist, CBT-1(Registered Trademark), Evaluating Pgp Inhibition in Tumors and Normal Tissues
Brief Title: Paclitaxel and CBT-1(Registered Trademark) to Treat Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan Bates, Dr. Susan Bates, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080035; 08-C-0035; NCT00658424 (obsolete NCT alias)
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Results first posted 2012-02-06 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Cervical; Ovarian; Lung; Breast; Renal
Keywords: Pgp; Solid Tumors; Drug Resistance; Sestamibi; Cancer; Solid Tumor
MeSH Terms: conditions — Neoplasms | interventions — Paclitaxel; Technetium Tc 99m Sestamibi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paclitaxel and CBT-1 (Experimental)
  Interventions: Drug: paclitaxel; Drug: CBT-1(Registered Trademark); Radiation: Tc 99m sestamibi

INTERVENTIONS:
Drug: paclitaxel — Paclitaxel 135 mg/m^2 intravenously on day 6 over 180 minutes. Cycles are repeated every 21 days.
  Other Names: Taxol; Onxal
Drug: CBT-1(Registered Trademark) — CBT-1 500 mg/m^2 oral dose daily for 7 days in divided doses 3 times a day. Cycle days 1-7, repeated every 21 days. no antacids, H2 blocker, or gastric acid inhibiting agents will be administered within 4 hours before or after each daily dose.
Radiation: Tc 99m sestamibi — 20 mCI baseline scan day 0; 20 mCI scan on 6th day of CBT-1 administered.

SUMMARY:
Background:

* Some cancer cells have a large amount of a protein called P-glycoprotein, which can pump certain chemotherapy drugs out of their cells. This pump may be part of the reason why it is difficult to shrink some cancers with chemotherapy.
* In laboratory experiments, the drug CBT-1(Registered Trademark) blocked the P-glycoprotein pump, resulting in accumulation of higher amounts of chemotherapy inside the cancer cells, making the chemotherapy more effective.
* Paclitaxel is a cancer drug that has caused tumors to shrink in many types of cancers, including lung, ovarian, breast, renal, cervical and others.

Objectives:

* To determine whether CBT-1(Registered Trademark) can block the P-glycoprotein pump on cancer cells and whether it inhibits the action of the pump found in normal blood cells and liver tissue.
* To evaluate the effectiveness of combination therapy using CBT-1(Registered Trademark) and paclitaxel in treating solid tumors and to determine whether the two drugs together are more effective than paclitaxel alone.

Eligibility:

-Patients over 18 years of age who have a solid tumor that cannot be treated successfully with standard treatments.

Design:

-Patients receive CBT-1(Registered Trademark) and paclitaxel in 21-day cycles. Treatment continues for two cycles after all the cancer is gone, or until it is decided to surgically remove some or all of the remaining cancer, or until the cancer has grown to the point where it defined as progressive disease.

For each cycle, patients take CBT-1(Registered Trademark) by mouth in three divided doses daily for 7 days. On day 6, paclitaxel is given through a vein over 3 hours.

Blood tests are done before starting CBT-1(Registered Trademark) and repeated periodically throughout treatment.

Imaging studies computed tomography or magnetic resonance imaging (CT or MRI) are done every two cycles. In addition, for the first cycle only, patients undergo imaging of tumors and normal tissue with a 99mTc-sestamibi radionuclide scan before and after administration of CBT-1(Registered Trademark). This scan helps show how well the P-glycoprotein pump is being blocked by the treatment.

DETAILED DESCRIPTION:
Background:

This is a pharmacodynamic study aimed at evaluating the efficacy of CBT-1(Registered Trademark) as a modulator of Pgp-mediated drug efflux in patient tumors and normal tissues. The study will build on over a decade of experience with 99mTc-sestamibi imaging and rhodamine accumulation and efflux in normal circulating CD56 plus cells as surrogates for Pgp function. CBA Research, Inc., has carried out Phase I and II testing of CBT-1(Registered Trademark) as a drug resistance reversal agent, but has not yet confirmed that the inhibitor is able to block drug efflux.

Objectives:

Evaluate the impact of CBT-1(Registered Trademark) on the hepatic accumulation and retention of 99mTc-sestamibi in patients with relapsed or refractory solid tumor malignancies.

Evaluate the impact of CBT-1(Registered Trademark) on P-glycoprotein-mediated efflux from CD56 plus peripheral mononuclear cells.

Eligibility:

Patients over 18 years of age who have histologic confirmation of relapsed/refractory cancer, following at least once standard treatment regimen, for whom there is no known standard therapy option capable of extending life expectancy. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 2 or better, and have hematologic, renal, hepatic, and metabolic parameters suggestive of adequate organ function.

Design:

Patients will be treated according to CBA Research Phase II trial of CBT-1 and Taxol. Patients will begin protocol treatment with orally administered CBT-1(Registered Trademark) in two or three divided doses daily for 7 days. On day 6, 135 mg/m^2 paclitaxel will be administered by intravenous infusion over 3 hours. Prior to the initiation of CBT-1(Registered Trademark), and on Day 6, patients will undergo blood sampling for the rhodamine assay in CD56 plus circulating mononuclear cells. In addition, patients will undergo imaging of tumors and normal tissue with the 99mTc-sestamibi radionuclide scan. These two assays have shown convincing inhibition of Pgp-mediated drug efflux in past studies with Pgp inhibitors such as tariquidar and valspodar. Twelve patients are planned for enrollment to this study, which is powered to determine a difference between the control scan and the post-treatment scan but not to compare CBT-1(Registered Trademark) with previous inhibitors tested in the intramural program.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must fulfill all of the following criteria to be eligible for study admission:

1. Age greater than 18 years.
2. Histologic or cytologic confirmation at National Cancer Institute (NCI) Laboratory of Pathology, of recurrent or refractory, or advanced metastatic cancer of the gastrointestinal tract, breast, Taxol (Trademark) naive breast cancer, small cell lung, ovarian, prostate, head and neck, multiple myeloma, non-small cell lung cancer, Taxol (Trademark) naive non-small cell lung cancer.
3. Performance status of Eastern Cooperative Oncology Group (ECOG) 0-2.
4. Life expectancy of 3 months or greater.
5. Patient must have adequate hematologic, renal, hepatic, and metabolic functions as defined: platelet count greater than 100,000 /mL, absolute granulocyte count (AGC) greater than 1500/mL, serum creatinine less than 2.0 mg/dl (or if greater than 2.0, a measured 24 hour creatinine clearance greater than 50 mL/min), serum glutamic oxaloacetic transaminase (SGOT) 4 times institutional upper limit of normal, bilirubin 2.0 mg/dl, prothrombin time (PT) less than 1.5 times institutional upper limit of normal, partial thromboplastin time (PTT) less than 1.5 times institutional upper limit of normal, calcium less than 5.3mEq/L, albumin greater than 2.0 g/dl.
6. Electrocardiogram (EKG) showing, at most, minor abnormalities that in the judgment of the protocol chairman would not compromise the patient's ability to tolerate therapy.
7. Patients must be greater than 4 weeks from prior radiation or chemotherapy; greater than 2 weeks from hormonal or immunotherapy; greater than 4 weeks from prior experimental therapy; greater than 6 weeks from mitomycin; and greater than 8 weeks from prior UCN01 treatment. Patients receiving dexamethasone as a pretreatment for anaphylactic reactions to Taxol (Trademark) or the cremophor vehicle will not be excluded from this study.
8. No serious intercurrent medical illness or serious infection that requires parenteral antibiotics.
9. Measurable disease by radiographic means or physical examination.
10. Willingness to sign a written informed consent.
11. Patients must agree to an effective method of contraception for the study (abstinence, hormonal or barrier method of birth control, or condom) for the study and 30 days after completion of protocol.

EXCLUSION CRITERIA:

The following patient populations are not eligible for study:

1. Women of childbearing potential and potentially fertile men will be excluded unless using an effective contraception (ie. a barrier intrauterine device (IUD), birth control pill, or condom), during the treatment. Women who are pregnant or nursing will also be excluded.
2. Patients with significant intercurrent disease.
3. Human Immunodeficiencey virus (HIV) seropositive patients. Note: There may be an impact of CBT-1 on the pharmacokinetics of the drugs used in the therapy of HIV.
4. Ongoing serious infections that require parenteral antibiotics.
5. Patients with significant central nervous system (CNS) disease, including a history of seizures within the last 3 months or psychiatric history which would impair the ability to give informed consent or prevent compliance with protocol requirements.
6. Patients must not be eligible for surgery, or radiotherapy that is of known benefit to them, in terms of extension of survival. Patients with tumors sensitive to potentially curative chemotherapy must have failed such chemotherapy. Patients who have received radiation therapy may participate in this study one week after the conclusion of radiation therapy provided that the lesion being irradiated is not one that is being used to assess the efficacy of CBT-1 plus Taxol.
7. History of significant coronary artery disease, cardiac arrhythmias requiring treatment, or history of other cardiac disease that in the judgment of the investigators, would compromise the patient's ability to tolerate the therapy.
8. Patients with active bleeding due to peptic ulcer disease.
9. History of anaphylactic reactions to paclitaxel or cremophor despite adequate premedication.
10. Clinically significant bleeding disorders.
11. Patients with solid organ allografts.
12. Patients on daily gastric acid secretion inhibitors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Bates, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Kelly RJ, Robey RW, Chen CC, Draper D, Luchenko V, Barnett D, Oldham RK, Caluag Z, Frye AR, Steinberg SM, Fojo T, Bates SE. A pharmacodynamic study of the P-glycoprotein antagonist CBT-1(R) in combination with paclitaxel in solid tumors. Oncologist. 2012;17(4):512. doi: 10.1634/theoncologist.2012-0080. Epub 2012 Mar 13. PMID 22416063
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2008-C-0035.html
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: US FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks
- See also: RECIST Criteria — http://ctep.cancer.gov/protocolDevelopment/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel and CBT-1 to Treat Solid Tumors: Patients will be treated with oral CBT-1 at a dose of 500 mg/m^2 daily for 7 days in divided doses and repeated every 21 days for 7 days beginning with cycle 1 of each cycle provided cycles are not delayed.
  Paclitaxel will be 135 mg/m^2 intravenously on day 6 over 180 minutes. Cycles are repeated every 21 days provided there is no delay, and will be administered on day 6 of each cycle.
Period: Overall Study
Arm/Group | Paclitaxel and CBT-1 to Treat Solid Tumors
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel and CBT-1 to Treat Solid Tumors
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 60.79 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 11
  Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent Increase in Sestamibi Retention in the Liver as a Measure of P-glycoprotein Inhibition
Description: An area under the concentration curve (AUC) was calculated for 99mTc counts over the liver, lungs, and heart. An equation was applied to determine the increase in sestamibi in the liver: [(AUCpost - AUC baseline)/(AUC baseline)] x 100.
Time Frame: sestamibi scanning was performed on day 0 and day 6, allowing scans to be performed pre and post CBT-1 administration
Population: As planned imaging data from 10 pts were analyzed.
Measure: Median (Full Range); unit: percent increase sestamibi retention
Arm/Group | Paclitaxel and CBT-1 to Treat Solid Tumors
Number analyzed (Participants) | 10
percent increase sestamibi retention | 71.9 [34.7 to 100.8]

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 18 months
Measure: Number; unit: Participants
Arm/Group | Paclitaxel and CBT-1 to Treat Solid Tumors
Number analyzed (Participants) | 12
Participants | 12

3. Secondary Outcome: Percent Inhibition of Rhodamine Efflux From CD56+Cells Post Treatment
Description: Rhodamine 123 was added to whole blood obtained before and after CBT-1. The blood was incubated, layered on lymphocyte separation medium and centrifuged. Peripheral blood mononuclear cells(PBMCs)were isolated, washed and incubated in rhodamine-free medium with or without valspodar. Cells were washed and incubated in phycoerythrin-labeled anti-CD56 antibody or negative control antibody. Rhodamine 123 fluorescence was assessed in CD56+cells with or without valspodar and a 60 min efflux period,continuing the cells without or with valspodar to generate Efflux and PSC/Efflux histograms.
Time Frame: Rhodamine efflux was performed on blood drawn prior to CBT-1 ingestion and after 6 days of dosing.
Population: Rhodamine 123 fluorescence was assessed in CD56+cells after a 30 min loading period with or without exogenously added valspodar and a 60 min efflux period followed, continuing the cells with or without exogenous valspodar to generate Efflux and PSC/Efflux histograms. Percent decrease in difference between these histograms is reported.
Measure: Mean (Full Range); unit: Percent inhibition of rhodamine efflux
Arm/Group | Paclitaxel and CBT-1 to Treat Solid Tumors
Number analyzed (Participants) | 12
Percent inhibition of rhodamine efflux | 78 [51 to 100]

4. Secondary Outcome: Number of Participants Who Had an Overall Response
Description: Response is determined by the Response Evaluation Criteria in Solid Tumors (RECIST) Criteria. Complete response (CR)-disappearance of all target lesions, Partial response (PR)-at least a 30% decrease in the sum of the longest diameter(LD)of target lesions, stable disease (SD) - neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
  See the Protocol Link module for further details about the RECIST Criteria.
Time Frame: Baseline to progression
Measure: Number; unit: participants with response
Arm/Group | Paclitaxel and CBT-1 to Treat Solid Tumors
Number analyzed (Participants) | 12
participants with response | 2

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Paclitaxel and CBT-1 to Treat Solid Tumors
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel and CBT-1 to Treat Solid Tumors (N=12)
Infection (pneumonia)with normal absolute neutrophil count (ANC) (Infections and infestations) | 1 (1)
Other: SVC (Superior vena cava) Syndrome (Vascular disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel and CBT-1 to Treat Solid Tumors (N=12)
ALKALINE PHOSPHATASE (Investigations) | 6 (8)
ALLERGIC REACTION (Immune system disorders) | 1 (1)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 2 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 3 (3)
ALT/SGPT (Investigations) | 5 (10)
ANOREXIA (Metabolism and nutrition disorders) | 6 (9)
AST/SGOT (Investigations) | 8 (12)
ATAXIA (Nervous system disorders) | 3 (4)
BICARBONATE, SERUM LOW (Investigations) | 2 (3)
BILIRUBIN (Investigations) | 4 (5)
BLURRED VISION (Eye disorders) | 1 (1)
CONFUSION (Psychiatric disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 4 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (5)
CREATININE (Investigations) | 1 (3)
DIARRHEA (Gastrointestinal disorders) | 9 (16)
DISTENTION (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (3)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 8 (9)
EDEMA, H&N (General disorders) | 2 (2)
EDEMA, LIMB (General disorders) | 3 (3)
FATIGUE (General disorders) | 10 (17)
FEVER (General disorders) | 3 (3)
FLUSHING (Vascular disorders) | 1 (1)
HEARTBURN (Gastrointestinal disorders) | 3 (5)
HEMOGLOBIN (Infections and infestations) | 12 (25)
HEMOGLOBINURIA (Renal and urinary disorders) | 1 (1)
HEMORRHAGE-GI, UPPER GI NOS (Gastrointestinal disorders) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 12 (28)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 3 (3)
HYPERURICEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 12 (17)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (5)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 7 (8)
HYPONATREMIA (Metabolism and nutrition disorders) | 8 (11)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 6 (10)
HYPOTENSION (Vascular disorders) | 3 (3)
HYPOTHYROIDISM (Endocrine disorders) | 1 (1)
INFECTION, URINARY TRACT NOS (Infections and infestations) | 1 (1)
INR (Investigations) | 1 (1)
LEUKOCYTES (Investigations) | 9 (14)
LYMPHOPENIA (Investigations) | 2 (2)
MOOD ALTERATION-ANXIETY (Psychiatric disorders) | 2 (2)
MUCOSITIS (CLINICAL EXAM), ORAL CAVITY (Gastrointestinal disorders) | 2 (2)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 10 (14)
NEUROPATHY-CRANIAL: CN-V MOTOR-JAW MUSCLES; SENSORY-FACIAL (Nervous system disorders) | 1 (1)
NEUROPATHY-SENSORY (Nervous system disorders) | 5 (5)
NEUTROPHILS (Investigations) | 8 (12)
OTHER: DYSURIA (Renal and urinary disorders) | 1 (1)
OTHER: INFECTION NOS (Infections and infestations) | 2 (2)
OTHER: LDH (Investigations) | 4 (4)
OTHER: PERFORATION NOS (Injury, poisoning and procedural complications) | 1 (1)
OTHER: PULMONARY STENOSIS NOS (Cardiac disorders) | 2 (2)
OTHER: RUQ PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN, THROAT/PHARYNX/LARYNX (Gastrointestinal disorders) | 1 (1)
PAIN NOS (General disorders) | 2 (2)
PAIN, ABD NOS (Gastrointestinal disorders) | 6 (8)
PAIN, BACK (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN, CHEST/THORAX NOS (Cardiac disorders) | 4 (4)
PAIN, HEAD/HEADACHE (Nervous system disorders) | 1 (1)
PAIN, JOINT (Musculoskeletal and connective tissue disorders) | 6 (10)
PAIN, MUSCLE (Musculoskeletal and connective tissue disorders) | 3 (4)
PAIN, RECTUM (Gastrointestinal disorders) | 1 (1)
PAIN, TUMOR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
PLATELETS (Investigations) | 5 (9)
PROTEINURIA (Renal and urinary disorders) | 6 (7)
PRURITIS (Skin and subcutaneous tissue disorders) | 1 (1)
PTT (Investigations) | 1 (1)
RIGORS/CHILLS (General disorders) | 2 (2)
TASTE ALTERATION (Gastrointestinal disorders) | 2 (2)
URINARY RETENTION (Renal and urinary disorders) | 2 (2)
VOICE CHANGES (Respiratory, thoracic and mediastinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 9 (12)
PLEURAL EFFUSION (Cardiac disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
MOOD ALTERATION, DEPRESSION (Psychiatric disorders) | 1 (1)
OTHER: LYMPHEDEMA (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No